CLINICAL TRIAL: NCT03901833
Title: Telemedicine Breastfeeding Support Following Late Preterm Delivery: A Randomized Controlled Trial
Brief Title: LIFT: Telemedicine Breastfeeding Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1382496
Record Dates: First submitted 2019-03-27; First posted 2019-04-03 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Support (Experimental): Weekly telemedicine breastfeeding support visits for four weeks, delivered via telemedicine
  Interventions: Behavioral: Telemedicine Support
- Control (Placebo Comparator): Standard of care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Telemedicine Support — Telemedicine intervention
  Arms: Telemedicine Support
Other: Standard of Care — Standard of Care
  Arms: Control

SUMMARY:
The central hypothesis guiding this project is that tailored breastfeeding support, that leverages easily accessible telemedicine technologies, can improve breastfeeding outcomes among late preterm dyads. The long-term goals of this project are to improve maternal and child health and reduce health disparities by designing and implementing evidence-based interventions to improve breastfeeding outcomes for this challenging patient population. This study seeks to identify lactation support practices that improve breastfeeding duration and to test the effect of telemedicine breastfeeding support on breastfeeding duration, among the nearly one in ten mothers who deliver late preterm (34-37 6/7 weeks), as this subpopulation of mothers faces the highest rates of premature breastfeeding cessation

ELIGIBILITY:
Inclusion Criteria:

* maternal age 18-49 years
* late preterm delivery (34-37 6/7 weeks)
* enrollment up to 1 week postpartum
* breastfeeding initiated
* access to a smartphone, tablet, or laptop computer in their home

Exclusion Criteria:

* incarceration
* inability to communicate in English
* infant with medical condition compromising breastfeeding (e.g. cleft lip and/or palate).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Experience | One month post-enrollment
  Mean score on a modified, 16-item Interactive Telehealth Satisfaction Scale >48 (corresponding to better than neutral on a 5 point Likert scale, 16 questions).

SECONDARY OUTCOMES:
Time to cessation | Monthly up to 12 months
  Time to breastfeeding cessation (assessed via monthly surveys as no to infant receiving any breast milk in last 24 hours)
Exclusive breastfeeding cessation | Monthly up to 12 months
  Time to exclusive breastfeeding cessation (assessed via monthly surveys, defined by initiation of formula, water, juice, other liquids, or solid foods)
Breastfeeding at 3 months | 3 months
  Proportion of infants breastfeeding at 3 months (assessed via 24 hour recall from infant's mother)
Exclusive breastfeeding | 3 months
  Proportion of infants breastfeeding without supplementation with other food or liquids at 3 months (assessed via 24 hour recall from infant's mother)
Individual satisfaction questions | 1 month post enrollment
  Mean satisfaction on each Interactive Telehealth Satisfaction Scale question

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kair, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California-Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/the-lift-study-telemedicine-breastfeeding-support-612908/